CLINICAL TRIAL: NCT07196280
Title: Protective Effect of 5-Alpha Reductase Inhibitors on Atherosclerotic Cardiovascular Disease in Populations With BPH: Evidence From UK Biobank Cohort and Chinese Single Center Database Studies
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Qing Yuan, Professor, Chinese PLA General Hospital
Other Study IDs: S2022-700-02
Record Dates: First submitted 2025-09-03; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Atherosclerotic Cardiovascular Disease (ASCVD); Benign Prostatic Hypertrophy (BPH)
MeSH Terms: conditions — Atherosclerosis; Prostatic Hyperplasia | interventions — 5-alpha Reductase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: 5-Alpha Reductase Inhibitors — Building on prior studies, drug exposure was defined as receiving 5-ARIs on at least two separate occasions, with an interval of no more than 180 days between prescriptions. Based on exposure status, the cohort was stratified into two groups.

SUMMARY:
To assess the impact of 5-alpha reductase inhibitors (5-ARIs) on the incidence of atherosclerotic cardiovascular disease (ASCVD) in patients with benign prostatic hyperplasia (BPH).

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with BPH or users of 5-ARIs

Exclusion Criteria:

* individuals who had cancer prior to the start of follow-up and those with pre-existing ASCVD

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population was derived from the UK Biobank (UKB). Detailed descriptions of the UKB have been published previously.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Atherosclerotic Cardiovascular Disease | Started taking 5α-reductase inhibitors until December 1, 2022
  While both CVD and ASCVD are composite disease categories, CVD encompasses a broader range of cardiovascular and cerebrovascular conditions. To ensure homogeneity in disease classification, we focused on ASCVD, which primarily refers to atherosclerosis-related cardiovascular and cerebrovascular diseases, including ischemic heart disease (IHD) and cerebrovascular disease (CeVD)

IPD SHARING:
Plan to Share IPD: No